CLINICAL TRIAL: NCT04412291
Title: A Multi-center, Randomized, Open-label Study in Patients With COVID-19 and Respiratory Distress Not Requiring Mechanical Ventilation, to Compare Standard-of-care With Anakinra and Tocilizumab Treatment The Immunomodulation-CoV Assessment (ImmCoVA) Study
Brief Title: A Study in Patients With COVID-19 and Respiratory Distress Not Requiring Mechanical Ventilation, to Compare Standard-of-care With Anakinra and Tocilizumab Treatment The Immunomodulation-CoV Assessment (ImmCoVA) Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jonas Sundén-Cullberg, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001748-24
Record Dates: First submitted 2020-06-01; First posted 2020-06-02 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Covid-19
Keywords: Coronavirus 2; SARS-CoV-2; Anakinra; Tocilizumab
MeSH Terms: conditions — COVID-19 | interventions — Steroids; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard-of-care Treatment (SOC) (Active Comparator): SOC according to local recommendations at the Karolinska University Hospital:
  Oxygen supplementation so to achieve SpO2>93%. Thrombosis prophylaxis (Fragmin or Innohep or Klexane or new oral anticoagulants incl. dabigatran, apixaban or rivaroxaban).
  Steroids (Betapred)
  Interventions: Drug: Standard-of-care treatment
- Anakinra + SOC (Active Comparator): Anakinra: A total dose of 400mg per day (divided in 4 doses of 100 mg iv every 6 hours) for 7 days.
  SOC according to local recommendations at the Karolinska University Hospital. Oxygen supplementation so to achieve SpO2>93%. Thrombosis prophylaxis (Fragmin or Innohep) Steroids (Betapred) Prophylactic broad spectrum antibiotics for seven days..
  Interventions: Drug: Anakinra Prefilled Syringe; Drug: Standard-of-care treatment
- Tocilizumab + SOC. (Active Comparator): Tocilizumab: 8mg/kg for a single infusion iv up to max 800 mg. If no clinical response is obtained, another dose of 8mg/kg may be administered after earliest 2 days SOC according to local recommendations at the Karolinska University Hospital. Oxygen supplementation so to achieve SpO2>93%. Thrombosis prophylaxis (Fragmin or Innohep) Steroids (Betapred) Prophylactic broad spectrum antibiotics for seven days.
  Interventions: Drug: Tocilizumab Prefilled Syringe; Drug: Standard-of-care treatment

INTERVENTIONS:
Drug: Anakinra Prefilled Syringe — A total dose of 400mg per day (divided in 4 doses of 100 mg iv every 6 hours) for 7 days.
  Arms: Anakinra + SOC
Drug: Tocilizumab Prefilled Syringe — 8mg/kg for a single infusion iv up to max 800 mg. If no clinical response is obtained, another dose of 8mg/kg may be administered after earliest 2 days after inclusion with the following condition: The clinical symptoms are worsened (as assessed by decreasing PaO2/FiO2 and/or need of increased ventilatory support such as NIV, HFNC or mechanical ventilation).
  Arms: Tocilizumab + SOC.
Drug: Standard-of-care treatment — SOC according to local recommendations at the Karolinska University Hospital. Oxygen supplementation so to achieve SpO2>93%. Thrombosis prophylaxis (Fragmin or Innohep and Klexane® or new oral anticoagulants including dabigatran, apixaban or rivaroxaban).
  Steroids (Betapred 6 mg po) Broad spectrum antibiotics (only in arm B and C)
  Other Names: Oxygen supplementation; Thrombosis prophylaxis; Steroids; Antibiotics

SUMMARY:
The study is designed as a randomized, controlled, multi-center open-label trial to compare standard-of-care (SOC) treatment with SOC + anakinra or SOC + tocilizumab treatment in hospitalized adult subjects who are diagnosed with severe COVID 19.

Arm A: Standard-of-care Treatment (SOC) Arm B: Anakinra + SOC Arm C: Tocilizumab + SOC.

All subjects will be treated with standard-of-care treatment. Arms B and C will also receive broad spectrum antibiotics initiated before or latest 24 hours after initiation of treatment with study drug.

The primary follow-up period of the study is 29 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay < 7 days prior to screening
3. SARS-CoV-2 infection with duration at least 7 days (i e may be included on day 7) as determined by onset of symptoms (defined as day 1)
4. 5 liters/minute of Oxygen for at least 8 hours to maintain SpO2 at ≥93%. A shorter duration is also accepted if presentation is acute, and the patient needs more than 10 liters/minute of Oxygen, or high flow nasal cannula or non-invasive ventilation, to maintain SpO2 at ≥93%..
5. CRP > 70 mg/L with no non-SARS-Cov2 infections. Values measured up to 48 hours before inclusion are accepted.
6. Ferritin > 500 µg/L Values measured up to 48 hours before inclusion are accepted.
7. At least two points on a scale of 0-3 where 1 point is awarded for each value of; lymphocytes < 1x 10(9)/L; D-dimer ≥ 0.5 mg/L and; Lactate Dehydrogenase ≥ 8 microkatal/L. The values do not have to be concurrently positive and may be up to 3 days old at inclusion.
8. Ability to provide informed consent signed by study patient
9. Willingness and ability to comply with study-related procedures/assessments
10. In fertile females, willing to comply with effective contraceptive methods for up to 3 months after last dose of study drug. These may include surgical sterilization of patient or partner, intrauterine device or condoms. Gestagen-only birth control pills (mini-pills), which do not increase the risk of deep venous thrombosis, may also be used. Non-fertile woman is defined as more than 12 months of amenorrhea without an alternative medical cause or, in case of ambiguities, an FSH level in the postmenopausal range.

Exclusion Criteria:

1. Pregnancy or breast feeding.
2. Ongoing or completed mechanical ventilation.
3. In the opinion of the investigator, unlikely to survive for >48 hours from screening.
4. In the opinion of the investigator, expected overall survival due to other comorbidities less than 3 months.
5. Severe renal dysfunction eGFR < 30 ml/min.
6. Medical history including chronic liver disease with inflammation, fibrosis or cirrhosis including underlying diseases such as alcoholic liver disease, non-alcoholic fatty liver disease, chronic viral hepatitis, alcoholic liver disease, autoimmune liver disease, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, cholangitis, or carcinoma.
7. Uncontrolled hypertension Systolic BP >180 mm Hg, Diastolic BP > 110 mm Hg.
8. History of hypersensitivity to the study drugs
9. Presence of any of the following abnormal laboratory values at screening: absolute neutrophil count (ANC) less than 2 x 109/L, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 5 x upper limit of normal (ULN), platelets <100 x 109/L
10. Treatment with anakinra, anti-IL 6, anti-IL-6R antagonists, Janus kinase inhibitors (JAKi) in the past 30 days or plans to receive during the study period
11. Current treatment with conventional synthetic disease-modifying antirheumatic drugs (DMARDs)/immunosuppressive agents
12. Use of chronic oral corticosteroids for a non-COVID-19-related condition in a dose higher than prednisone 10 mg or equivalent per day. Ongoing acute treatment for COVID-19 with any peroral or iv steroid is permitted for up to five days before inclusion. Chronic or acute treatment with inhaled steroids is also permitted
13. History of, or current autoimmune or inflammatory systemic or localized disease(s) other than rheumatoid arthritis
14. Acute systemic infection; verified by blood cultures systemic bacterial infection, systemic fungi-infection or prosthesis-related infection
15. History of stem-cell or solid organ transplantation
16. Known active tuberculosis (TB), history of incompletely treated TB, suspected or known extrapulmonary TB, suspected or known systemic bacterial or fungal infections
17. Diagnosis of, or suspicion of HIV infection, acute hepatitis A and/or chronic hepatitis B and/or C
18. Previous history of gastrointestinal ulceration or diverticulitis.
19. Patients who have received immunosuppressive antibody therapy within the past 3 months, including intravenous immunoglobulin or plans to receive during the study period
20. Participation in any clinical research study evaluating an investigational product (IP) or therapy within 3 months and less than 5 half-lives of IP prior to the screening visit. The use of remdesivir is permitted.
21. Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Time to recovery | Day 1 through Day 29
  Day of recovery is defined as the first day on which the subject satisfies one of the following three categories from the ordinal scale:1) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care 1; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 3) Not hospitalized, no limitations on activities.
  1 LMWH-injections (Fragmin, Innohep) do not count as medical care

SECONDARY OUTCOMES:
Mortality | Up to day 29
Number of Days on mechanical ventilation | Up to day 29
Number of days of supplemental oxygen use | Up to day 29
Number of patients requiring initiation of mechanical ventilation | Up to day 29
Time to improvement in oxygenation for at least 48 hours | Up to day 29
  Definition of improvement in oxygenation: Increase in SpO2/FiO2 of 50 or greater compared to the nadir SpO2/FiO2
Mean change in the 8-point ordinal scale | Up to day 15
  8-point Ordinal Scale:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO;
  3. Hospitalized, on non-invasive ventilation or high flow nasal cannula;
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen;
  8. Not hospitalized
Proportion of patients on level e-h on the 8-point ordinal scale at day 15 | Day 15
  8-point Ordinal Scale:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO;
  3. Hospitalized, on non-invasive ventilation or high flow nasal cannula;
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen;
  8. Not hospitalized
Time to improvement in one category from baseline using the 8-point ordinal scale | Up to day 29
  8-point Ordinal Scale:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO;
  3. Hospitalized, on non-invasive ventilation or high flow nasal cannula;
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen;
  8. Not hospitalized
Mean change in Sequential organ failure assessment score (SOFA) | Up to day 15
Time to resolution of fever for at least 48 hours by clinical severity | Up to day 29
  Defined as ≤36.6°C (axilla), ≤37.2°C (oral) or ≤37.8°C (rectal or tympanic)
Time to improvement of three points from baseline in National Early Warning Score 2 (NEWS2) scoring system | Up to day 29
  NEWS2 consists of: Physiological Parameters: Respiration rate (per minute), SpO2 Scale 1 (%), SpO2 Scale 2 (%), Use of air or oxygen, Systolic blood pressure (mmHg), Pulse (per minute), Consciousness, Temperature (°C)
Time to score of <2 maintained for 24 hours in NEWS2 scoring system (National Early Warning Score) | Up to day 29
  NEWS2 consists of: Physiological Parameters: Respiration rate (per minute), SpO2 Scale 1 (%), SpO2 Scale 2 (%), Use of Air or oxygen, Systolic blood pressure (mmHg), Pulse (per minute), Consciousness, Temperature (°C)
Mean change in NEWS2 scoring system (National Early Warning Score) | Up to day 15
Number of days with fever. | Up to day 29
  Based on highest measured daily body temperature. Defined as >36.6°C (axilla), >37.2°C (oral) or >37.8°C (rectal or tympanic
Number of days of resting respiratory rate >24 breaths/min | Up to day 29
  Based on highest respiratory rate measured between 06.00 and 09.00 each day
Time to saturation ≥94% on room air | Up to day 29
Cumulative dose of steroids; equivalent to betamethasone dosage (mg) | From start of steroid treatment for Covid-19 up to day 29
Cumulative dose of steroids during the study; equivalent to betamethasone dosage (mg) | From day 1 up to day 29
Incidence of serious adverse events | Up to day 60
Incidence of severe or life-threatening bacterial, invasive fungal, or opportunistic infection | Up to day 29
Incidence of severe or life-threatening bacterial, invasive fungal, or opportunistic infection in patients with grade 4 neutropenia | Up to day 60
Incidence of hypersensitivity reactions | Up to day 29
Incidence of infusion reactions | Up to day 29
Number of ventilator free days in the first 28 days | Baseline to day 29
Number of patients requiring non-invasive ventilation | Up to day 29
Number of patients requiring the use of high flow nasal cannula | Up to day 29
Number of patients requiring Extracorporeal membrane oxygenation (ECMO) | Up to day 29
Number of patients that have been admitted into an intensive care unit (ICU) | Up to day 29
Number of patients that have been admitted into a High Dependency Unit ("Intermediärvårdsavdelning") | Up to day 29
Number of days admitted into a High Dependency Unit ("Intermediärvårdsavdelning") or intensive care unit (ICU) [ | Up to day 29
Number of days of hospitalization in survivors | Up to day 29
Number of patients discharged to institution other than normal domicile. | Up to day 60
Number of deaths due to any cause | Up to day 60

CONTACTS AND LOCATIONS:
Overall Officials: jonas Sundén-Cullberg, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Sunden-Cullberg J, Chen P, Habel H, Skorup P, Janols H, Rasmuson J, Niward K, Ostholm Balkhed A, Chatzidionysiou K, Asgeirsson H, Blennow O, Parke A, Svensson AK, Muvva JR, Ljunggren HG; Karolinska KI/K COVID-19 Treatment Working Group; Horne AC, Aden U, Henter JI, Sonnerborg A, Vesterbacka J, Nowak P, Lampa J. Anakinra or tocilizumab in patients admitted to hospital with severe covid-19 at high risk of deterioration (IMMCoVA): A randomized, controlled, open-label trial. PLoS One. 2023 Dec 29;18(12):e0295838. doi: 10.1371/journal.pone.0295838. eCollection 2023. PMID 38157348